CLINICAL TRIAL: NCT00089648
Title: A Phase 2 Study Of SU011248 In The Treatment Of Patients With Bevacizumab-Refractory Metastatic Renal Cell Carcinoma
Brief Title: SU011248 In The Treatment Of Patients With Bevacizumab (Avastin)-Refractory Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181039
Record Dates: First submitted 2004-08-09; First posted 2004-08-11 (Estimated); Results first posted 2009-12-21 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — 50 mg orally daily for 4 weeks followed by 2 weeks off treatment for approximately 1 year or until disease progression/unacceptable toxicity; after completion of 1 year, pts with clinical benefit can continue the study treatment in a separate continuation protocol
  Other Names: SUTENT, SU011248,

SUMMARY:
The purpose of this study is to test whether sunitinib (SU011248) has activity and is safe in patients with renal cell carcinoma (RCC) who have failed prior therapy with bevacizumab (Avastin) -based treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven renal cell carcinoma of clear cell histology with metastases
* Evidence of measurable disease
* Radiographic evidence of disease progression during or within 3 months of completion of bevacizumab-based treatment
* Prior radical or partial nephrectomy

Exclusion Criteria:

* Prior treatment with any other anti-angiogenic therapy other than bevacizumab
* Prior systemic treatment for RCC > 2 regimens
* History of or known brain metastases
* Serious acute or chronic illness or recent history of significant cardiac abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2004-12; Primary Completion 2007-01 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - Pfizer Investigational Site, Duarte, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181039&StudyName=SU011248%20In%20The%20Treatment%20Of%20Patients%20With%20Bevacizumab%20%28Avastin%29-Refractory%20Metastatic%20Renal%20Cell%20Carcinoma%20%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: 50 milligram/day for 4 consecutive weeks followed by a 2-week off-treatment period (6-week treatment cycle).
Period: Overall Study
Arm/Group | Sunitinib
Started | 61
Completed | 20
Not Completed | 41
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 33

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 61
Age, Customized [Number; unit: participants]
  < 65 years | 43
  > = 65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Overall Confirmed Objective Disease Response According to the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Objective disease response = subjects with confirmed complete response (CR) or partial response (PR) according to RECIST. A CR was defined as the disappearance of all target lesions. A PR was defined as a ≥ 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: 4 week treatment cycles up to 1 year in absence of withdrawal criteria requiring discontinuation including 28 day post study follow up
Population: Intent-to-treat (ITT)=all subjects enrolled in the study that received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 61
participants | 14
Statistical Analysis 1: Comparison: Sunitinib; Test type: Superiority or Other; Objective Response Rate (ORR) (percent) = 23.0, 95% CI [13.2 to 35.5] — ORR=proportion of subjects with confirmed CR or PR, relative to total number of subjects who received at least 1 dose of study medication, were refractory to bevacizumab, had a baseline disease assessment and had the correct histological cancer type

2. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP was defined as the time from the date of first dose of study medication to the date of the first documentation of tumor progression. If tumor progression data included more than 1 date, the first date was used. TTP (in weeks) was calculated as (first event date minus first dose date +1)/7. Kaplan-Meier method was used.
Time Frame: as for outcome 1
Population: ITT. 20 subjects were censored.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 61
weeks | 30.4 [18.3 to 36.7]

3. Secondary Outcome: Duration of Response (DR)
Description: DR was defined as the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or to death due to to any cause that occurred within 28 days after the last dose of study medication, whichever occurred first. If tumor progression data included more than 1 date, the first date was used. DR was only calculated for the subgroup of subjects with a confirmed objective response. DR was calculated as [the end date for DR minus first CR or PR that was subsequently confirmed +1]/7. Kaplan-Meier method was used.
Time Frame: as for outcome 1
Population: ITT subjects (i.e, all subjects enrolled in the study that received at least 1 dose of study medication) who had a confirmed CR or PR. 14 subjects who had a response were analyzed for DR.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 61
weeks | 36.1 [25.0 to 999]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from start of study treatment to date of death due to any cause. OS (in weeks) was calculated as [date of death minus first dose date +1]/7. For a subject not expiring, the OS time was censored on the last date of known contact that they were known to be alive. Subjects lacking data beyond the day of the first dose had their OS times censored at 1 day. Kaplan-Meier method was used.
Time Frame: as for outcome 1
Population: ITT
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 61
weeks | 47.1 [36.9 to 69.7]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from start of study medication to first documentation of objective tumor progression or to death due to any cause that occurred on treatment including within 28 days after the last dose of study medication, whichever occurred first. If tumor progression data included more than 1 date, the first date was used. PFS (in weeks) was calculated as (first event date minus first dose date +1)/7. Kaplan-Meier method was used.
Time Frame: as for outcome 1
Population: ITT. 20 subjects were censored.
Measure: Median (Full Range); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 61
weeks | 30.4 [18.3 to 36.7]

6. Secondary Outcome: Trough Plasma Concentrations (Cmin) of Sunitinib
Time Frame: Day 28 of Cycle 1 to Cycle 4
Population: ITT
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 59
ng/mL
  Cycle 1, Day 28 (n=20) | 52.05 [29.80 to 91.40]
  Cycle 2, Day 28 (n=23) | 43.50 [8.69 to 93.00]
  Cycle 3, Day 28 (n=10) | 46.10 [24.80 to 72.00]
  Cycle 4, Day 28 (n=16) | 44.90 [13.10 to 103.00]

7. Secondary Outcome: Trough Plasma Concentrations (Cmin) of SU012662
Time Frame: Day 28 of Cycle 1 to Cycle 4
Population: ITT
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 59
ng/mL
  Cycle 1, Day 28 (n=20) | 30.50 [14.10 to 64.00]
  Cycle 2, Day 28 (n=23) | 21.40 [5.51 to 55.20]
  Cycle 3, Day 28 (n=10) | 22.10 [8.49 to 40.70]
  Cycle 4, Day 28 (n=16) | 23.75 [11.40 to 47.80]

8. Secondary Outcome: Trough Plasma Concentrations (Cmin) of Total Drug (Sunitinib + SU012662)
Time Frame: Day 28 of Cycle 1 to Cycle 4
Population: ITT
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 59
ng/mL
  Cycle 1, Day 28 (n=20) | 85.40 [43.90 to 141.70]
  Cycle 2, Day 28 (n=23) | 66.60 [18.32 to 129.40]
  Cycle 3, Day 28 (n=10) | 68.40 [41.29 to 106.10]
  Cycle 4, Day 28 (n=16) | 68.15 [29.20 to 126.00]

9. Secondary Outcome: Plasma Concentration of Vascular Endothelial Growth Factor-A (VEGF-A)
Description: Plasma concentrations of VEGF-A that may be associated with tumor proliferation or angiogenesis collected from a subset of subjects were analyzed by ELISA analysis. Samples below the limit of quantitation and samples with insufficient volume available were excluded.
Time Frame: Cycle 1 (Days 1, 14, and 28), Cycle 2 (Day 1)
Population: ITT
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 61
pg/mL
  Cycle 1, Day 1 (Baseline) (n=59) | 567.4 [57 to 3692]
  Cycle 1, Day 14 (n=57) | 1320.6 [104.5 to 4751]
  Cycle 1, Day 28 (n=55) | 1212.3 [105.2 to 6137]
  Cycle 2, Day 1 (n=54) | 316.2 [56.9 to 1724]

10. Secondary Outcome: Plasma Concentration of Soluble VEGF Receptor-3 (sVEGFR-3)
Description: Plasma concentrations of sVEGFR-3 that may be associated with tumor proliferation or angiogenesis collected from a subset of subjects were analyzed by ELISA analysis. Samples below the limit of quantitation and samples with insufficient volume available were excluded.
Time Frame: Cycle 1 (Days 1, 14, and 28), Cycle 2 (Day 1)
Population: ITT
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 61
pg/mL
  Cycle 1, Day 1 (Baseline) (n=54) | 54170.4 [21300 to 202900]
  Cycle 1, Day 14 (n=32) | 37747.0 [21500 to 122900]
  Cycle 1, Day 28 (n=22) | 46891.0 [22700 to 109700]
  Cycle 2, Day 1 (n=46) | 51280.0 [21700 to 122900]

11. Secondary Outcome: Plasma Concentration of Placental Growth Factor (PlGF)
Description: Plasma concentrations of PlGF that may be associated with tumor proliferation or angiogenesis collected from a subset of subjects were analyzed by ELISA analysis. Samples below the limit of quantitation and samples with insufficient volume available were excluded.
Time Frame: Cycle 1 (Days 1, 14, and 28)
Population: ITT
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 61
pg/mL
  Cycle 1, Day 1 (Baseline) (n=37) | 55.0 [24.4 to 257]
  Cycle 1, Day 14 (n=58) | 146.1 [44.8 to 408]
  Cycle 1, Day 28 (n=53) | 137.9 [28.2 to 490]

12. Secondary Outcome: Plasma Concentration of VEGF-C
Description: Plasma concentrations of VEGF-C that may be associated with tumor proliferation or angiogenesis collected from a subset of subjects were analyzed by ELISA analysis. Samples below the limit of quantitation and samples with insufficient volume available were excluded.
Time Frame: Cycle 1 (Days 1, 14, and 28)
Population: ITT
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 61
pg/mL
  Cycle 1, Day 1 (Baseline) (n=57) | 833.0 [332 to 3167]
  Cycle 1, Day 14 (n=57) | 688.0 [284.5 to 1353]
  Cycle 1, Day 28 (n=54) | 566.5 [213 to 1391]

13. Secondary Outcome: Plasma Concentration of Soluble VEGF Receptor-2(sVEGFR-2)
Description: Plasma concentrations of sVEGFR-2 that may be associated with tumor proliferation or angiogenesis collected from a subset of subjects were to have been analyzed by ELISA analysis; however, no data were collected.
Time Frame: 1 year
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 30/61
Other Adverse Events (participants affected / at risk) | 60/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=61)
Anaemia (Blood and lymphatic system disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 5
Fatigue (General disorders) | 4
Pyrexia (General disorders) | 2
Chest pain (General disorders) | 1
Generalised oedema (General disorders) | 1
Oedema (General disorders) | 1
Pain (General disorders) | 1
Diverticulitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Wound infection (Infections and infestations) | 2
Abdominal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=61)
Anaemia (Blood and lymphatic system disorders) | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Hypothyroidism (Endocrine disorders) | 14
Lacrimation increased (Eye disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 10
Cheilitis (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 25
Diarrhoea (Gastrointestinal disorders) | 42
Dry mouth (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 20
Eructation (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10
Glossodynia (Gastrointestinal disorders) | 4
Haemorrhoids (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 37
Stomatitis (Gastrointestinal disorders) | 28
Vomiting (Gastrointestinal disorders) | 29
Chest pain (General disorders) | 8
Chills (General disorders) | 12
Fatigue (General disorders) | 54
Mucosal inflammation (General disorders) | 21
Oedema peripheral (General disorders) | 20
Pain (General disorders) | 5
Pyrexia (General disorders) | 13
Sinusitis (Infections and infestations) | 8
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 10
Excoriation (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 8
Blood creatinine increased (Investigations) | 9
Blood glucose increased (Investigations) | 4
Blood phosphorus decreased (Investigations) | 4
Blood uric acid increased (Investigations) | 4
Ejection fraction decreased (Investigations) | 7
Haemoglobin decreased (Investigations) | 5
Lipase increased (Investigations) | 5
Neutrophil count decreased (Investigations) | 8
Platelet count decreased (Investigations) | 5
Weight decreased (Investigations) | 11
Weight increased (Investigations) | 5
White blood cell count decreased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 37
Dehydration (Metabolism and nutrition disorders) | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hyponatraemia (Metabolism and nutrition disorders) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 14
Flank pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20
Dizziness (Nervous system disorders) | 12
Dysgeusia (Nervous system disorders) | 34
Headache (Nervous system disorders) | 14
Peripheral sensory neuropathy (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 6
Confusional state (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 20
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 12
Exfoliative rash (Skin and subcutaneous tissue disorders) | 5
Hair colour changes (Skin and subcutaneous tissue disorders) | 8
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 22
Periorbital oedema (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 12
Skin discolouration (Skin and subcutaneous tissue disorders) | 24
Skin reaction (Skin and subcutaneous tissue disorders) | 11
Hypertension (Vascular disorders) | 20
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.